CLINICAL TRIAL: NCT03821792
Title: A Phase 2 Course Determining Study for Men With Hormone-Naïve Metastatic Prostate Cancer (HNMPCa)
Brief Title: Abiraterone Acetate, Prednisone, and Apalutamide in Treating Patients With Hormone-Naive Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0533; NCI-2018-03599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0533 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Prostate Carcinoma Metastatic in the Bone; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abiraterone acetate, prednisone, apalutamide) (Experimental): Patient receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily. Cycles repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies how well abiraterone acetate, prednisone, and apalutamide work in treating patients with hormone-naive prostate cancer that has spread to other places in the body. Androgen can cause the growth of prostate cancer cells. Antihormone therapy, such as abiraterone acetate and apalutamide may lessen the amount of androgen made by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if a baseline molecular-pathologic androgen receptor response (AR-response) signature predicts efficacy to abiraterone plus apalutamide in patients with hormone-naive metastatic prostate cancer (HNMPCa).

SECONDARY OBJECTIVES:

I. Evaluate the efficacy of abiraterone acetate plus apalutamide in patients with HNMPCa.

II. Evaluate the safety of abiraterone acetate plus apalutamide in patients with HNMPCa.

III. Explore the relationship between molecular markers and clinical efficacy outcomes.

OUTLINE:

Patient receive abiraterone acetate orally (PO) daily, prednisone PO twice daily (BID), and apalutamide PO daily. Cycles repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* At least 2 of the 3 following high-risk prognostic factors:

  * Gleason score of >= 8
  * Presence of 3 or more lesions on bone scan
  * Presence of measurable visceral (excluding lymph node disease) metastasis on computed tomography (CT) or magnetic resonance imaging (MRI) (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Hemoglobin >= 9.0 g/dL independent of transfusion and/or growth factors within 3 months prior to enrollment
* Platelet count >= 100,000/uL independent of transfusion and/or growth factors within 3 months prior to enrollment
* Serum albumin >= 3.0 g/dL
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Calculated creatinine clearance (Cockcroft-Gault equation) >= 45 mL/min
* Serum potassium >= 3.5 mEg/L
* Serum magnesium >= 1.6 mg/dL
* Serum bilirubin < 1.5 x institutional upper limit of normal (IULN) (except for patients with known Gilbert's disease if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible)
* Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x IULN for patients without liver metastases. (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible. For patients with liver metastases AST or ALT < 4 x IULN is allowed)
* Able to swallow study drugs whole as a tablet/capsule
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug
* Patients must agree to tissue collection for correlative studies at the specified time points

Exclusion Criteria:

* Small cell prostate cancer
* Treatment within 28 days of cycle 1 day 1: Any prior pharmacotherapy, radiation therapy, or surgery for metastatic prostate cancer. The following exceptions are permitted:

  * Up to 3 months of antiandrogen therapy (ADT) with LHRH agonists or antagonists or orchiectomy with or without concurrent anti-androgens prior to cycle 1 day 1. Anti-androgens (flutamide, bicalutamide or nilutamide) for subjects receiving an LHRH agonist must be discontinued within 2 weeks of cycle 1 day 1, or subjects may have one course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease (e.g., impending cord compression or obstructive symptoms) if it was administered at least 28 days prior to cycle 1 day 1. All adverse events associated with these procedures must be resolved at least to grade 1 by cycle 1 day 1, or
* Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone daily. Use of inhaled, intranasal, intra-articular and topical steroids are acceptable, as is a short course (i.e. =< 1 day) of corticosteroids to prevent a reaction to the intravenous (IV) contrast used for CT scans
* Active infection (requiring oral or IV antibiotics or antiviral therapy) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* A malignancy (other than the one treated in this study) which required radiotherapy or systemic treatment within the past 5 years, or has a >= 30% probability of recurrence within 24 months (except for non-melanoma skin cancer or Ta urothelial carcinomas)
* Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 170 or diastolic pressures above 110 despite anti-hypertensive therapy. Note that this is NOT a criterion related to particular blood pressure (BP) results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes. (For example doctor's visit related stress i.e. "white coat syndrome")
* Prolonged corrected QT interval by Fridericia's formula (QTcF) interval on pre-entry electrocardiogram (>= 450 msec)
* Known active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de pointes), New York Heart Association class III-IV heart disease or cardiac ejection fraction measurement of < 40% at baseline
* Patients who have had a history of illness which put them at current risk for bowel perforation such as acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis
* Baseline moderate and severe hepatic impairment (Child Pugh class B & C)
* Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
* Gastrointestinal disorder affecting absorption
* Untreated symptomatic spinal cord compression
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2026-10-11 (Estimated); Study Completion 2026-10-11 (Estimated)

PRIMARY OUTCOMES:
Time on treatment | Up to 6 months
  Calculated as the time from start of protocol treatment

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from starting treatment until progression, assessed up to 6 months
  Median PFS and 95% confidence interval will be presented for all patients and by the androgen receptor molecular-pathologic responsiveness signature.
Incidence of adverse events | Up to 6 months
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Efficacy assessed | Up to 6 months
  prostate specific antigen, bone specific alkaline phosphatase, and urine n-telopeptides
Expression of candidate markers | Up to 6 months
  Candidate markers for different biologic domains by immunohistochemistry, mass spectrometry (for steroid metabolome) and genomic profiling. Markers will encompass bone remodeling (e.g. integrin signaling), steroid metabolome (e.g. glucocorticoid receptor) and tumor immunoprofile (e.g. PD-1, PDL-1).
Overall survival | up to 6 months
  Time from start of protocol treatment until death or last contact

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M Anderson Cancer Center — http://www.mdanderson.org